CLINICAL TRIAL: NCT04007328
Title: To Assess the Role of Sphingosine-1-phosphate in the Pathobiology of Pneumonia: Generate a New Strategy for Treatment of Severe Community-acquired Pneumonia
Brief Title: Sphingosine-1-phosphate and Pneumonia
Acronym: SOPN
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201812054
Record Dates: First submitted 2019-04-23; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Pneumonia, Bacterial
Keywords: sphingosine-1-phosphate; corticosteroids adjuvant therapy
MeSH Terms: conditions — Pneumonia, Bacterial | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- methylprednisolone (Experimental): 20 mg of methylprednisolone IV Q12H for 5 days
  Interventions: Drug: Methylprednisolone Sodium Succinate
- Placebo (Placebo Comparator): normal saline IV Q12H for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone Sodium Succinate — methylprednisolone vial
  Arms: methylprednisolone
Drug: Placebo — Normal saline manufactured to mimic methylprednisolone vial
  Arms: Placebo

SUMMARY:
Pneumonia is a major infectious cause of death worldwide and imposes a considerable burden on healthcare resources. Sphingosine-1-phosphate (S1P) is a bioactive sphingolipid and involved in many physiological processes including immune responses and endothelial barrier integrity. In term of endothelial barrier integrity, S1P plays a crucial role in protecting lungs from pulmonary leak and lung injury. Because of the involvement in lung injury, S1P could be the potential biomarker of pneumonia. Recently, our pilot study suggested that patients with CAP have significantly higher plasma S1P levels than healthy individuals. Interestingly, our observational study also showed significantly elevated S1P level in the patients who were treated with methylprednisolone during the hospitalization. Based on the above evidence, we hypothesize that S1P plays an important role in the pathobiology of pneumonia. Moreover, S1P is not only a useful biomarker for diagnosis of CAP, but also can be an indicator for using corticosteroids adjuvant therapy.

DETAILED DESCRIPTION:
Lower respiratory tract infections are the most frequent infectious cause of death worldwide[1] and impose a considerable burden on healthcare resources. Sphingosine-1-phosphate (S1P) is a bioactive sphingolipid and has both extracellular and intracellular effects in mammalian cells[2-5]. S1P is involved in many physiological processes including immune responses and endothelial barrier integrity[6-9]. In the context of endothelial barrier integrity, S1P plays a crucial role in protecting the lungs from the pulmonary leak and lung injury. [10-13] Previous research suggests that, at low concentrations, S1P signaling through S1PR1 is crucial for enhancing endothelial barrier function. [13,14] The S1P induces actin polymerization and results in the spreading of endothelial cells, which fill the intercellular gaps. Also, the S1P signaling can stabilize the endothelial cell-cell junctions, such as adherens junction and tight junction. [15-17] Both actin-dependent outward spreading of endothelial cells and cell junction stabilization enhance the endothelial barrier function. However, S1P at higher concentration (> 5 µM) causes endothelial barrier disruption through binding of S1PR2[13]. Thus, exact maintenance of physiologic S1P concentrations and homeostasis of S1PRs and S1P synthesis and degradation seem to be crucial for the preservation of lung endothelial barrier integrity, particularly in inflammatory lung diseases.

Because of the involvement in lung injury and endothelial barrier function, S1P may be a potential biomarker of pneumonia. Moreover, a recent study proposed that targeting the S1P/S1P receptor 2-signaling pathway in the lung may provide a novel therapeutic perspective in pneumonia for the prevention of acute lung injury [18]. Recently, our pilot study suggests that the patients with CAP (N= 137) have significantly higher plasma S1P levels than controls (N= 78). Further, the S1P levels, but not CRP, were found to be inversely correlated with PSI score, CURB-65 score and hospital length of stay (LOS) in patients with CAP. Our initial findings suggest that plasma S1P is a potential biomarker for predicting prognosis in CAP.

Although corticosteroids adjuvant therapy for CAP is still controversial, a recent meta-analysis study showed that corticosteroids adjuvant therapy in patients with the severe CAP could reduce the rate of in-hospital mortality and reduce the length of hospital stay[19]. Recently, the long-standing dogma of cytokine repression by the glucocorticoid was challenged. Vettorazzi et al. proposed a new mechanism of glucocorticoid action. They suggested that increased circulating sphingosine 1-phosphate levels resulting from the induction of sphingosine kinase 1 (SphK1) by glucocorticoids were essential for the inhibition of pulmonary inﬂammation[20]. Interestingly, our observational study also showed significantly elevated S1P levels in patients who were treated with methylprednisolone during hospitalization.

Several studies have suggested that S1P can enhance pulmonary endothelial cell barrier function, suggesting that higher S1P levels could be potentially beneficial. Hence, the patients, who are unable to produce sufficient S1P, might have a poor prognosis. However, in most of the studies, CAP was not considered as a disease model, and those results were based on cell lines and mouse models. Therefore, further clinical studies focusing on the role of S1P in the pathophysiology of pneumonia is needed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms suggestive community-acquired pneumonia and pneumonia severe index (PSI) > 90, Age 18 years or older and Written informed consent obtained

Exclusion Criteria:

* Presence of severe immunosuppression (HIV infection, use of immunosuppressants), malignancy, pregnancy or breastfeeding, patient with uncontrol diabetes, current use of antibiotics or corticosteroids, any likely infection other than CAP, or pneumonia that developed within 3 days after hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Mortality | up to 4 months
  In hospital mortality

SECONDARY OUTCOMES:
ICU Admission | up to 4 months
  If the patient has any Intensive Care Unit (ICU) Admission?
Length of ICU stay | up to 4 months
  Length of ICU stay (day)
length of hospital stay | up to 4 months
  length of hospital stay (day)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Wang Hsu, MD, Principal Investigator — Wan Fang Hospital
Locations (1):
- Wan Fang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lozano R, Naghavi M, Foreman K, Lim S, Shibuya K, Aboyans V, Abraham J, Adair T, Aggarwal R, Ahn SY, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Barker-Collo S, Bartels DH, Bell ML, Benjamin EJ, Bennett D, Bhalla K, Bikbov B, Bin Abdulhak A, Birbeck G, Blyth F, Bolliger I, Boufous S, Bucello C, Burch M, Burney P, Carapetis J, Chen H, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, De Leo D, Degenhardt L, Delossantos A, Denenberg J, Des Jarlais DC, Dharmaratne SD, Dorsey ER, Driscoll T, Duber H, Ebel B, Erwin PJ, Espindola P, Ezzati M, Feigin V, Flaxman AD, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabriel SE, Gakidou E, Gaspari F, Gillum RF, Gonzalez-Medina D, Halasa YA, Haring D, Harrison JE, Havmoeller R, Hay RJ, Hoen B, Hotez PJ, Hoy D, Jacobsen KH, James SL, Jasrasaria R, Jayaraman S, Johns N, Karthikeyan G, Kassebaum N, Keren A, Khoo JP, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lipnick M, Lipshultz SE, Ohno SL, Mabweijano J, MacIntyre MF, Mallinger L, March L, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGrath J, Mensah GA, Merriman TR, Michaud C, Miller M, Miller TR, Mock C, Mocumbi AO, Mokdad AA, Moran A, Mulholland K, Nair MN, Naldi L, Narayan KM, Nasseri K, Norman P, O'Donnell M, Omer SB, Ortblad K, Osborne R, Ozgediz D, Pahari B, Pandian JD, Rivero AP, Padilla RP, Perez-Ruiz F, Perico N, Phillips D, Pierce K, Pope CA 3rd, Porrini E, Pourmalek F, Raju M, Ranganathan D, Rehm JT, Rein DB, Remuzzi G, Rivara FP, Roberts T, De Leon FR, Rosenfeld LC, Rushton L, Sacco RL, Salomon JA, Sampson U, Sanman E, Schwebel DC, Segui-Gomez M, Shepard DS, Singh D, Singleton J, Sliwa K, Smith E, Steer A, Taylor JA, Thomas B, Tleyjeh IM, Towbin JA, Truelsen T, Undurraga EA, Venketasubramanian N, Vijayakumar L, Vos T, Wagner GR, Wang M, Wang W, Watt K, Weinstock MA, Weintraub R, Wilkinson JD, Woolf AD, Wulf S, Yeh PH, Yip P, Zabetian A, Zheng ZJ, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2095-128. doi: 10.1016/S0140-6736(12)61728-0. PMID 23245604
- [Background] Rosen H, Goetzl EJ. Sphingosine 1-phosphate and its receptors: an autocrine and paracrine network. Nat Rev Immunol. 2005 Jul;5(7):560-70. doi: 10.1038/nri1650. PMID 15999095
- [Background] Anliker B, Chun J. Cell surface receptors in lysophospholipid signaling. Semin Cell Dev Biol. 2004 Oct;15(5):457-65. doi: 10.1016/j.semcdb.2004.05.005. PMID 15271291
- [Background] Meyer zu Heringdorf D, Liliom K, Schaefer M, Danneberg K, Jaggar JH, Tigyi G, Jakobs KH. Photolysis of intracellular caged sphingosine-1-phosphate causes Ca2+ mobilization independently of G-protein-coupled receptors. FEBS Lett. 2003 Nov 20;554(3):443-9. doi: 10.1016/s0014-5793(03)01219-5. PMID 14623109
- [Background] Usatyuk PV, He D, Bindokas V, Gorshkova IA, Berdyshev EV, Garcia JG, Natarajan V. Photolysis of caged sphingosine-1-phosphate induces barrier enhancement and intracellular activation of lung endothelial cell signaling pathways. Am J Physiol Lung Cell Mol Physiol. 2011 Jun;300(6):L840-50. doi: 10.1152/ajplung.00404.2010. Epub 2011 Apr 8. PMID 21478254
- [Background] Pappu R, Schwab SR, Cornelissen I, Pereira JP, Regard JB, Xu Y, Camerer E, Zheng YW, Huang Y, Cyster JG, Coughlin SR. Promotion of lymphocyte egress into blood and lymph by distinct sources of sphingosine-1-phosphate. Science. 2007 Apr 13;316(5822):295-8. doi: 10.1126/science.1139221. Epub 2007 Mar 15. PMID 17363629
- [Background] Rivera J, Proia RL, Olivera A. The alliance of sphingosine-1-phosphate and its receptors in immunity. Nat Rev Immunol. 2008 Oct;8(10):753-63. doi: 10.1038/nri2400. PMID 18787560
- [Background] Schuchardt M, Tolle M, Prufer J, van der Giet M. Pharmacological relevance and potential of sphingosine 1-phosphate in the vascular system. Br J Pharmacol. 2011 Jul;163(6):1140-62. doi: 10.1111/j.1476-5381.2011.01260.x. PMID 21309759
- [Background] Xiong Y, Hla T. S1P control of endothelial integrity. Curr Top Microbiol Immunol. 2014;378:85-105. doi: 10.1007/978-3-319-05879-5_4. PMID 24728594
- [Background] Dudek SM, Jacobson JR, Chiang ET, Birukov KG, Wang P, Zhan X, Garcia JG. Pulmonary endothelial cell barrier enhancement by sphingosine 1-phosphate: roles for cortactin and myosin light chain kinase. J Biol Chem. 2004 Jun 4;279(23):24692-700. doi: 10.1074/jbc.M313969200. Epub 2004 Mar 31. PMID 15056655
- [Background] McVerry BJ, Peng X, Hassoun PM, Sammani S, Simon BA, Garcia JG. Sphingosine 1-phosphate reduces vascular leak in murine and canine models of acute lung injury. Am J Respir Crit Care Med. 2004 Nov 1;170(9):987-93. doi: 10.1164/rccm.200405-684OC. Epub 2004 Jul 28. PMID 15282202
- [Background] Peng X, Hassoun PM, Sammani S, McVerry BJ, Burne MJ, Rabb H, Pearse D, Tuder RM, Garcia JG. Protective effects of sphingosine 1-phosphate in murine endotoxin-induced inflammatory lung injury. Am J Respir Crit Care Med. 2004 Jun 1;169(11):1245-51. doi: 10.1164/rccm.200309-1258OC. Epub 2004 Mar 12. PMID 15020292
- [Background] Sammani S, Moreno-Vinasco L, Mirzapoiazova T, Singleton PA, Chiang ET, Evenoski CL, Wang T, Mathew B, Husain A, Moitra J, Sun X, Nunez L, Jacobson JR, Dudek SM, Natarajan V, Garcia JG. Differential effects of sphingosine 1-phosphate receptors on airway and vascular barrier function in the murine lung. Am J Respir Cell Mol Biol. 2010 Oct;43(4):394-402. doi: 10.1165/rcmb.2009-0223OC. Epub 2009 Sep 11. PMID 19749179
- [Background] Li X, Stankovic M, Bonder CS, Hahn CN, Parsons M, Pitson SM, Xia P, Proia RL, Vadas MA, Gamble JR. Basal and angiopoietin-1-mediated endothelial permeability is regulated by sphingosine kinase-1. Blood. 2008 Apr 1;111(7):3489-97. doi: 10.1182/blood-2007-05-092148. Epub 2008 Jan 16. PMID 18199826
- [Background] Camerer E, Regard JB, Cornelissen I, Srinivasan Y, Duong DN, Palmer D, Pham TH, Wong JS, Pappu R, Coughlin SR. Sphingosine-1-phosphate in the plasma compartment regulates basal and inflammation-induced vascular leak in mice. J Clin Invest. 2009 Jul;119(7):1871-9. doi: 10.1172/jci38575. PMID 19603543
- [Background] Xu M, Waters CL, Hu C, Wysolmerski RB, Vincent PA, Minnear FL. Sphingosine 1-phosphate rapidly increases endothelial barrier function independently of VE-cadherin but requires cell spreading and Rho kinase. Am J Physiol Cell Physiol. 2007 Oct;293(4):C1309-18. doi: 10.1152/ajpcell.00014.2007. Epub 2007 Aug 1. PMID 17670896
- [Background] Arce FT, Whitlock JL, Birukova AA, Birukov KG, Arnsdorf MF, Lal R, Garcia JG, Dudek SM. Regulation of the micromechanical properties of pulmonary endothelium by S1P and thrombin: role of cortactin. Biophys J. 2008 Jul;95(2):886-94. doi: 10.1529/biophysj.107.127167. Epub 2008 Apr 11. PMID 18408039
- [Background] Gutbier B, Schonrock SM, Ehrler C, Haberberger R, Dietert K, Gruber AD, Kummer W, Michalick L, Kuebler WM, Hocke AC, Szymanski K, Letsiou E, Luth A, Schumacher F, Kleuser B, Mitchell TJ, Bertrams W, Schmeck B, Treue D, Klauschen F, Bauer TT, Tonnies M, Weissmann N, Hippenstiel S, Suttorp N, Witzenrath M; CAPNETZ Study Group. Sphingosine Kinase 1 Regulates Inflammation and Contributes to Acute Lung Injury in Pneumococcal Pneumonia via the Sphingosine-1-Phosphate Receptor 2. Crit Care Med. 2018 Mar;46(3):e258-e267. doi: 10.1097/CCM.0000000000002916. PMID 29298188
- [Background] Wu WF, Fang Q, He GJ. Efficacy of corticosteroid treatment for severe community-acquired pneumonia: A meta-analysis. Am J Emerg Med. 2018 Feb;36(2):179-184. doi: 10.1016/j.ajem.2017.07.050. Epub 2017 Jul 15. PMID 28756034
- [Background] Vettorazzi S, Bode C, Dejager L, Frappart L, Shelest E, Klassen C, Tasdogan A, Reichardt HM, Libert C, Schneider M, Weih F, Henriette Uhlenhaut N, David JP, Graler M, Kleiman A, Tuckermann JP. Glucocorticoids limit acute lung inflammation in concert with inflammatory stimuli by induction of SphK1. Nat Commun. 2015 Jul 17;6:7796. doi: 10.1038/ncomms8796. PMID 26183376